CLINICAL TRIAL: NCT01760720
Title: Methadone Maintenance Treatment (MMT) Care for HIV Prevention: A Randomized Controlled Trial (MMT2)
Brief Title: Methadone Maintenance Treatment (MMT) Care for HIV Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Li Li, PhD, Professor in Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA033130 (NIH)
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Stigma
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention): Standard care
- intervention (Experimental): The MMT CARE intervention has 3 session/modules: 1) MMT protocol and procedures, understanding stigma and its impact; 2) effective communication with clients, introducing motivational interviewing; 3) application of motivational interviewing, motivating clients for behavior change. The intervention contents reflect challenges faced by service providers working at MMT clinics and the impact of these challenges on their clients. Sessions will occur once a week for three weeks, with each session featuring a different set of themes and relevant activities. Each session will be 90-100 minutes long and will be conducted with a group of 5 to 7 providers.
  Interventions: Behavioral: MMT CARE

INTERVENTIONS:
Behavioral: MMT CARE
  Arms: intervention

SUMMARY:
Based on our previous success with the intervention pilot (R34MH083512), we conducted this randomized controlled trial (MMT CARE), which will integrate behavioral intervention components with a primarily pharmacological model of MMT. The intervention focuses on treatment adherence and effective outcomes by reducing stigmatizing attitudes and behaviors among service providers, enhancing their communication skills, and improving their interactions with and support of their clients' behavior changes. Our goal is to bring a contextual change to support a protective environment for clients' motivation and capacity in order to reduce their HIV risk. The findings could benefit not only China but also the global community by effectively combining interventions for controlling the HIV epidemic.

DETAILED DESCRIPTION:
Injecting drug use is the major mode of HIV transmission for 740,000 people living with HIV (PLH) in China. In response to this situation, China introduced methadone maintenance treatment (MMT) in 2004, which is now dispensed by 701 clinics serving 295,000 clients. Despite this impressive scale-up, China's MMT programs still face serious challenges, including high drop-out rates, a large number of clients who continue to use heroin during MMT, a gap between clients' needs and services availability, providers' lack of skills in counseling and education, and stigma linked to resistance to harm reduction. This study aims to address these challenges.

Based on our previous success with the intervention pilot (R34MH083512), we conducted this randomized controlled trial (MMT CARE), which will integrate behavioral intervention components with a primarily pharmacological model of MMT. The intervention focuses on treatment adherence and effective outcomes by reducing stigmatizing attitudes and behaviors among service providers, enhancing their communication skills, and improving their interactions with and support of their clients' behavior changes. Our goal is to bring a contextual change to support a protective environment for clients' motivation and capacity in order to reduce their HIV risk. The findings could benefit not only China but also the global community by effectively combining interventions for controlling the HIV epidemic.

The study will be implemented in Sichuan, Guangdong, Hunan, Shaanxi and Jiangsu provinces. A total of 68 MMT clinics will be randomly selected from the five provinces and randomized to either the intervention condition (MMT CARE group) or the control condition. From each selected clinic, we will recruit 6 service providers and 36 clients, totaling 408 service providers and 2,448 clients (204 service provider and 1,224 clients in each condition, respectively).

The Specific Aims of the study are as follows:

1. To examine whether providers in the intervention group, compared to providers in the control group, demonstrate improved adherence to MMT protocols, decreased prejudicial attitudes, increased interactions with clients, and increased communications with clients on risk reduction.
2. To examine whether MMT clients in the intervention group, compared to clients in the control group, demonstrate improved treatment adherence/retention, decreased concurrent drug use, increased motivation for behavior change, improved mental health, increased positive support, and reduced HIV risk behaviors.
3. To explore whether providers' improved outcomes are associated with improved client outcomes.

ELIGIBILITY:
Inclusion Criteria:

MMT clients

* Age 20 and above
* Currently enrolled in MMT at the participating clinics
* Informed consent Service providers
* Age 18 and above
* Currently working in the participating MMT clinics
* Informed consent

Exclusion Criteria:

MMT Clients

* Psychosis, neurological damage, as judged by an interviewer in consultation with a clinical supervisor
* Currently under criminal or civil charges
* Inability to give informed consent
* Anyone who does not meet the inclusion criteria

Service Providers

* Inability to give informed consent
* Anyone who does not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2866 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Client treatment retention | Change from baseline to 6-, 12-, 18- and 24-month follow up
  MMT retention will be measured by the treatment status (in treatment vs. drop out) at each follow-up point.

SECONDARY OUTCOMES:
Client's mental health | Change from baseline to 6-, 12-, 18- and 24-month follow up
  The Zung Depression Scale will be used to measure clients' depressive symptoms. Drug avoidance self-efficacy will be measured with selected questions from the Drug Avoidance Self-Efficacy Scale (DASES).
Provider attitudes toward and interaction with clients | Change from baseline to 6-, 12-, 18- and 24-month follow up
  Negative attitude toward drug users will be measured with questions adapted from the brief scale of attitude measurement developed by researchers at the National Centre for Education and Training on Addiction, Flinders University, Australia (2006). Provider-client interaction will be measured with 12 questions specifically developed for this study and tested in the pilot.

CONTACTS AND LOCATIONS:
Overall Officials: Zunyou Wu, PhD, Study Director — China CDC
Locations (1):
- China CDC, NCAIDS, Beijing, China

REFERENCES:
- [Derived] Li L, Liang LJ, Lin C, Feng N, Cao W, Wu Z. An intervention to improve provider-patient interaction at methadone maintenance treatment in China. J Subst Abuse Treat. 2019 Apr;99:149-155. doi: 10.1016/j.jsat.2019.01.022. Epub 2019 Feb 3. PMID 30797387